CLINICAL TRIAL: NCT04472949
Title: Thoracic Radiotherapy Plus Maintenance Durvalumab After First Line Carboplatin and Etoposide Plus Durvalumab in Extensive-stage Disease Small Cell Lung Cancer (ED-SCLC). A Multicenter Single Arm Open Label Phase II Trial.
Brief Title: Thoracic Radiotherapy Plus Maintenance Durvalumab After First Line Carboplatin and Etoposide Plus Durvalumab in Extensive-stage Disease Small Cell Lung Cancer (ED-SCLC).
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 15/19
Record Dates: First submitted 2020-07-10; First posted 2020-07-16 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Small Cell Lung Cancer; Lung Cancer
Keywords: small cell lung cancer; lung cancer; ED-SCLC; Thoracic radiotherapy; Durvalumab; extensive-stage disease small cell lung cancer; Prospective; multicenter; single-arm; phase II trial; open-label; Carboplatin; Etoposide
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — durvalumab; Carboplatin; Etoposide

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, open-label, single-arm, phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab & thoratic radiotherapy (Experimental): Patients will start with an induction phase (part 1). Patients with CR; PR or SD after the induction phase, will transfer to the maintenance phase (part 2). Patients with PD after the induction phase will transfer to the follow-up phase.
  Induction phase (part 1):
  Patients will receive durvalumab in combination with carboplatin and etoposide for 4 cycles of 21 days:
  Maintenance phase (part 2):
  Patients will receive durvalumab treatment up to PD or max. 2 years, i.e. 26 maintenance cycles, in combination with tRT:
  Follow up phase:
  Patients will be followed up for 24 months, every 8 weeks.
  Interventions: Drug: Durvalumab; Drug: carboplatin; Drug: etoposide; Radiation: Thoracic radiotherapy

INTERVENTIONS:
Drug: Durvalumab — Durvalumab: 1500 mg iv
  Other Names: MEDI4736
Drug: carboplatin — Carboplatin: AUC 5 mg/mL/min iv
Drug: etoposide — Etoposide: 100 mg/m2 iv
Radiation: Thoracic radiotherapy — Thoracic radiotherapy: 39 Gy in 13 fractions, starting 3-8 weeks after day 1 of last cycle of induction treatment, over 2.5 weeks Prophylactic cranial irradiation (PCI) is allowed but optional: according to local practice, starting 3-8 weeks after day 1 of last cycle of induction treatment Follow up phase Patients will be followed up for 24 months, every 8 weeks.

SUMMARY:
Standard of care for Extensive-Stage Disease (ED) Small Cell Lung Cancer (SCLC) as first-line treatment is 4 to 6 cycles of platinum based chemotherapy (carboplatin or cisplatin) in combination with etoposide. However, the outcome of the disease remains poor with a median overall survival of approximately 10 months, mainly caused by rapid development of drug resistance. The risk of intrathoracic recurrences can be reduced and an improved 2-year survival can be achieved with the addition of thoracic radiotherapy (tRT).

The main objective of the trial is to evaluate the efficacy of tRT combined with maintenance durvalumab in SCLC after chemoimmunotherapy. Secondary objective is to evaluate the safety of tRT combined with maintenance durvalumab in SCLC after chemo-immunotherapy.

For this trial durvalumab is the IMP. Patients will start with an induction phase (part 1): Patients will receive durvalumab in combination with carboplatin and etoposide for 4 cycles of 21 days.

Patients with CR; PR or SD after the induction phase, will transfer to the maintenance phase (part 2): Patients will receive durvalumab treatment up to PD or max. 2 years, i.e. 26 maintenance cycles, in combination with tRT.

Patients with PD after the induction phase will transfer to the follow-up phase: Patients will be followed up for 24 months, every 8 weeks.

DETAILED DESCRIPTION:
The prognosis of patients with advanced small cell lung cancer is poor. Despite chemotherapy and immunotherapy, median survival is only 12 months. The trial SAKK 15/19 is investigating whether thoracic radiotherapy and the administration of durvalumab can slow down the progression of the disease.

In patients with advanced small cell lung cancer, the standard therapy consists of 4-6 cycles of platinum-based chemotherapy plus etoposide with or without Atezolizumab. Nevertheless, the median overall survival of these patients is only 10-12 months, because resistance to the therapy usually develops rapidly.

Radiotherapy and maintenance therapy with Durvalumab to activate the immune system The risk of intrathoracic progression of small cell lung cancer can be reduced by additional thoracic radiotherapy. It is assumed that the radiation not only has a direct cytotoxic effect on the tumor cells, but also stimulates an antitumor immune response.

In the trial SAKK 15/19, it is being investigated whether the combination of the monoclonal anti-PD-L1 antibody durvalumab with thoracic radiotherapy in patients with advanced small cell lung cancer can cause an even stronger activation of the immune system with an improved antitumoral immune response. The trial therapy (thoracic radiotherapy + durvalumab) is based on chemo-immunotherapy with carboplatin, etoposide and durvalumab. The primary endpoint of the trial is the progression-free rate after 12 months, secondary endpoints include progression-free survival, median overall survival and objective response rate.

Which patients can participate? The trial is open to patients with advanced small-cell lung cancer who have either metastases (stage IV) or whose lung tumor volume is so large that radiation therapy with curative intent is not possible as a first-line therapy (stage III-IV). Patients who have already received systemic therapy or thoracic radiotherapy because of the small cell lung carcinoma cannot participate.

Conduct of the trial

Participation in the trial is carried out in three phases for patients:

* Induction therapy: Patients receive four cycles of chemo-immunotherapy with carboplatin, etoposide and durvalumab. One cycle lasts 21 days. In those patients who show a response or stable disease situation after completion of induction therapy, maintenance therapy follows. Maintenance therapy is not performed in patients whose disease has progressed further under induction therapy.
* Maintenance therapy: Thoracic radiotherapy for 2.5-3 weeks (13 fractions of 3 Gray each) and administration of Durvalumab every 28 days for a maximum of two years.
* Follow-up for two years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH-GCP E6(R2) regulations before registration and prior to any trial specific procedures
* Histologically or cytologically1 confirmed extensive disease stage IV SCLC (T any, N any, M1 a/b) or T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan (according to American Joint Committee on Cancer Stage (8th edition)
* Patients must be considered suitable to receive carboplatin with etoposide as 1st line treatment for the ED-SCLC
* Patients with brain metastases are also eligible provided they are asymptomatic or treated central nervous system metastases and meet the following criteria:

  * No ongoing requirement for corticosteroids at least 2 weeks prior to trial treatment
  * No leptomeningeal disease
* Patients with a prior malignancy other than SCLC and treated with curative intention are eligible, if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease at registration. Less than 2 years is acceptable for malignancies with low risk of recurrence and/or no late recurrence, after consultation with the Coordinating Investigator
* Measurable disease per RECIST v1.1
* Age ≥ 18 years
* WHO performance status 0-1
* Adequate pulmonary function: forced expiratory volume in one second FEV (1) ≥ 1.0 liter
* Adequate bone marrow function:

  * Absolute neutrophil count ≥ 1.5 x 109/L1
  * Platelet count ≥ 100 x 109/L
  * Hemoglobin ≥ 90 g/L
* Adequate hepatic function:

  * Total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN)
  * AST and/or ALT ≤ 2.5 x ULN (in patients with hepatic metastasis: AST and/or ALT ≤ 5.0 x ULN)
* Adequate renal function measured (by the CKD-EPI formula) or calculated creatinine clearance ≥ 45 mL/min (by the Cockcroft-Gault formula)
* Women of childbearing potential must use highly effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and until 90 days after the last dose of investigational drug. A negative serum pregnancy test performed within 7 days before registration is required for all women of childbearing potential
* Men agree not to donate sperm or to father a child during trial treatment and until 90 days after the last dose of investigational drug

Exclusion criteria:

* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 1 week prior to registration
* Prior chemotherapy treatment for ED-SCLC
* Any history of radiotherapy to the chest. Radiation therapy outside of the chest for palliative care (i.e., bone metastasis) is allowed but must be completed before first dose of -
* Prior systemic treatment including immune checkpoint inhibitors against SCLC
* Concomitant treatment within 30 days of registration with any other experimental drug and/or enrollment in another clinical trial
* Concomitant use of other anti-cancer drugs or radiotherapy. Except surgery for local pain control
* Severe or uncontrolled cardiovascular disease

  * Congestive heart failure NYHA III or IV;
  * Unstable angina pectoris
  * History of myocardial infarction within the last 3 months
  * Serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia)
  * Uncontrolled hypertension
* Uncontrolled or symptomatic hypercalcemia, i.e.

  * > 1.5 mmol/L ionized calcium
  * > 12 mg/dL or > 3 mmol/L corrected serum calcium
* Known interstitial lung disease
* Body weight ≤ 30 kg
* Major surgical procedure (defined by the investigator) within 28 days prior to the first dose of durvalumab or anticipation of need for a major surgical procedure during the course of the trial
* Known history of active primary immunodeficiency
* Known history of human immunodeficiency virus (HIV) or active chronic Hepatitis C or Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous antimicrobial treatment
* Known history of allogeneic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders including:

  * Inflammatory bowel disease (e.g., colitis or Crohn's disease)
  * Systemic lupus erythematosus
  * Wegener syndrome (granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.)
* Patients with eczema, psoriasis, lichen simplex chronicus are not permitted, except they are with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) and meet the following conditions:

  * Rash must cover less than 10% of body surface area
  * Disease is well controlled at baseline and only requires low potency topical steroids
  * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency, or oral steroids)
* Patients with a paraneoplastic syndrome (PNS) of autoimmune nature, requiring systemic treatment (systemic steroids or immunosuppressive agents) or has a clinical symptomatology suggesting worsening of PNS
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening thorax CT scan
* Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab
* Concomitant or prior use, i.e. within 14 days before the first dose of durvalumab, of immunosuppressive medication including immunosuppressant, such as methotrexate, azathioprine and tumor necrosis factor (TNF)-α blockers, with the exceptions of:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiological doses not to exceed 10 mg/day of prednisone or an equivalent corticosteroid
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) and premedication for chemotherapy
* Known hypersensitivity to the drugs used in this trial (carboplatin, etoposide, durvalumab)
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free rate (PFR) (RECIST v.1.1) | at 12 months after registration
  PFR (RECIST v.1.1) at 12 months after registration, defined by the Kaplan-Meier estimator for progression-free survival (RECIST v.1.1) at 12 months (+ 4 weeks as we allow 4 weeks delay in the tumor assessment at 12 months).

SECONDARY OUTCOMES:
Progression-free survival (PFS) (RECIST v.1.1) | From the date of registration until the date of progressive disease according to RECIST v1.1 or death, whichever occurs first, assessed up to 4 years after registration.
  PFS (RECIST v.1.1), defined as the time from registration until progression according to RECIST v1.1 or death from any cause, whichever occurs first. Patients without an event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of the last tumor assessment before the start of the new therapy, if any.
Progression-free survival (PFS) (RECIST v.1.1) outside the brain | From the date of registration until the date of progressive disease according to RECIST v1.1 or death, whichever occurs first, assessed up to 4 years after registration
  PFS (RECIST v.1.1) outside the brain, defined as progression-free survival, except that relapses in the brain will be censored.
Progression-free survival (RECIST v.1.1) after induction chemotherapy (PFS-IND) | From the date of completion of induction chemotherapy until the date of progressive disease according to RECIST v1.1 or death, whichever occurs first, assessed up to 4 years after registration
  PFS-IND defined as the time from completion of induction chemotherapy until progression according to RECIST v1.1 or death from any cause, whichever occurs first. Patients without an event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of the last tumor assessment before the start of the new therapy, if any. PFS-IND will only be analyzed in patients who had CR, PR or SD after induction chemotherapy and started radiotherapy maintenance.
Overall Survival (OS) | From the date of registration until the date of death, assessed up to 4 years after registration
  OS defined as the time from registration until death from any cause. Patients without an event at the time of analysis will be censored at the date they were last known to be alive.
Objective response rate (ORR) | From the date of registration until the date of progressive disease according to RECIST v1.1 or death, whichever occurs first, assessed up to 4 years after registration
  ORR defined as proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 during trial treatment.
Duration of response (DOR) | From the date of first CR or PR according to RECIST v1.1 until the date of progressive disease according to RECIST v1.1, relapse or death, whichever occurs first, assessed up to 4 years after registration
  DOR defined as time from the date when a patient first meets the criteria for CR or PR according to RECIST v1.1, until documented progression, relapse or death due to disease progression, whichever occurs first. Patients without an event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of the last tumor assessment before the start of the new therapy, if any. DOR will only be analyzed in patients achieving CR or PR during trial treatment.
Adverse events (AEs) | From the date of registration to 90 days after last trial treatment
  AEs assessed according to NCI CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Addeo, Prof, Study Chair — Hôpitaux Universitaires Genève
Locations (14):
- Switzerland (14):
  - Kantonsspital Aarau, Aarau
  - Universitaetsspital Basel, Basel
  - IOSI Ospedale Regionale di Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Hôpitaux Universitaires de Genève, Geneva
  - Klinik Hirslanden, Männedorf
  - Spital Männedorf, Männedorf
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital Thun, Thun
  - HFR Freiburg - Kantonsspital, Villars-sur-Glâne
  - Kantonsspital Winterthur, Winterthur
  - UniversitätsSpital Zürich, Zurich